CLINICAL TRIAL: NCT02404610
Title: Moderate Versus Deep Procedural Sedation With Propofol in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR 13-3746
Record Dates: First submitted 2014-10-20; First posted 2015-03-31 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Pain
Keywords: propofol; moderate procedural sedation; deep procedural sedation; memory; emergency department
MeSH Terms: conditions — Pain; Emergencies | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Procedural Sedation (Experimental): Subjects will undergo procedural sedation for an indicated urgent medical procedure with a target sedation level of moderate sedation. Moderate procedural sedation is a specific term referring to procedural sedation with a target depth of moderate.
  Interventions: Procedure: Moderate Procedural Sedation with a sedative medication.; Drug: propofol
- Deep Procedural Sedation (Experimental): Subjects will undergo procedural sedation for an indicated urgent medical procedure with a target sedation level of deep sedation. Deep procedural sedation is a specific term referring to procedural sedation with a target depth of deep.
  Interventions: Procedure: Deep Procedural Sedation with a sedative medication.; Drug: propofol

INTERVENTIONS:
Procedure: Moderate Procedural Sedation with a sedative medication. — procedural sedation with a target sedation depth of moderate. Moderate sedation is not a drug specific intervention, it is achieved with the use of a sedative or a combination of sedations and opioids.
  Arms: Moderate Procedural Sedation
Procedure: Deep Procedural Sedation with a sedative medication. — procedural sedation with a target sedation depth of deep. Deep sedation is not a drug specific intervention, it is achieved with the use of a sedative or a combination of sedations and opioids.
  Arms: Deep Procedural Sedation
Drug: propofol

SUMMARY:
This study is a clinical trial of moderate sedation versus deep sedation with propofol for procedural sedation in the Emergency Department. The purpose of this study is to compare the rate of amnesia and respiratory depression rate in patients who receive moderate sedation to those that receive deep sedation.

DETAILED DESCRIPTION:
Purpose: For the pilot phase, if the visual memory assessment test developed in this study can adequately assess periods of amnesia during the procedure, then it can be used for the phase of the study that randomizes patients to moderate or deep sedation. The purpose of the randomized phase is to compare the rate of amnesia and respiratory depression in patients who receive moderate sedation to those that received deep sedation. The goal is to determine whether moderate sedation could provide a safer sedation while still resulting in adequate amnesia of the procedure. Secondary goals would be to compare the duration of sedation, the success of the procedures for which the patient is sedated, procedural difficulty, the rate of hypotension and other adverse events, and the patient perception of the quality of the sedation (pain or recall of procedure).

Background: Adequate pain control and alleviation of anxiety improves quality of care and patient satisfaction. Numerous studies have found that procedural sedation (PS) in the ED is safe, and when properly administered, the incidence of reported complications, including clinically significant respiratory depression, is rare. Procedural sedation is used for procedures such as fracture reduction, dislocation reduction, cardioversion, incision and drainage, and chest tube placement. Propofol is an anesthetic agent frequently used for PS in the Emergency Department (ED) and produces sedation, hypnosis, and amnesia, but lacks analgesic properties. In studies conducted at Hennepin County Medical Center (HCMC), we have found that patients are unable to recall whether or not they experienced pain during the procedure when sedated with propofol. However, there is the possibility that certain parts of the procedure can be later recalled by the patient. If extensive parts of the procedure can be recalled, then this is not an effective sedation. Previous studies of memory during sedation at HCMC have used verbal prompts only, but research has shown that people can more readily remember images. Images may provide a more sensitive way to determine the degree of amnesia during sedation.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing procedural sedation with propofol in the emergency department

Exclusion Criteria:

* < 18 years old
* Pregnant
* Previous allergic reaction to propofol
* Prisoner
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-07; Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Schick, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Miner JR, Danahy M, Moch A, Biros M. Randomized clinical trial of etomidate versus propofol for procedural sedation in the emergency department. Ann Emerg Med. 2007 Jan;49(1):15-22. doi: 10.1016/j.annemergmed.2006.06.042. Epub 2006 Sep 25. PMID 16997421
- [Background] Miner JR, Biros M, Krieg S, Johnson C, Heegaard W, Plummer D. Randomized clinical trial of propofol versus methohexital for procedural sedation during fracture and dislocation reduction in the emergency department. Acad Emerg Med. 2003 Sep;10(9):931-7. doi: 10.1111/j.1553-2712.2003.tb00646.x. PMID 12957974
- [Background] Miner JR, Biros MH, Seigel T, Ross K. The utility of the bispectral index in procedural sedation with propofol in the emergency department. Acad Emerg Med. 2005 Mar;12(3):190-6. doi: 10.1197/j.aem.2004.10.004. PMID 15741580

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Procedural Sedation: Subjects will undergo procedural sedation for an indicated urgent medical procedure with a target sedation level of moderate sedation. Moderate procedural sedation is a specific term referring to procedural sedation with a target depth of moderate.
  Moderate Procedural Sedation with a sedative medication.: procedural sedation with a target sedation depth of moderate. Moderate sedation is not a drug specific intervention, it is achieved with the use of a sedative or a combination of sedations and opioids.
  propofol
- Deep Procedural Sedation: Subjects will undergo procedural sedation for an indicated urgent medical procedure with a target sedation level of deep sedation. Deep procedural sedation is a specific term referring to procedural sedation with a target depth of deep.
  Deep Procedural Sedation with a sedative medication.: procedural sedation with a target sedation depth of deep. Deep sedation is not a drug specific intervention, it is achieved with the use of a sedative or a combination of sedations and opioids.
  propofol
Period: Overall Study
Arm/Group | Moderate Procedural Sedation | Deep Procedural Sedation
Started | 54 | 53
Completed | 54 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Procedural Sedation | Deep Procedural Sedation | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 100
  >=65 years | 3 | 4 | 7
Age, Continuous [Median (Full Range); unit: years] | 41.5 [18 to 78] | 39 [20 to 73] | 40 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 24 | 28 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54 | 53 | 107

OUTCOME MEASURES:

1. Primary Outcome: Patients With Clinical Signs of Respiratory Depression or Sub Clinical Respiratory Depressions Measured by Capnography and Pulse Oximetry.
Description: adverse respiratory events measured using capnography, pulse oximetry, and airway maneuvers performed during the sedation procedure
Time Frame: From start of procedure until the patient has returned to baseline mental status after the conclusion of the sedation procedure, an expected average time of 30 minutes
Population: patients undergoing procedural sedation in the ED
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Procedural Sedation | Deep Procedural Sedation
Number analyzed (Participants) | 54 | 53
Participants | 22 | 21

ADVERSE EVENTS:
Time Frame: From 3 minutes prior to the start of the sedation encounter up until the time the patient regained their baseline mental status up to 24 hours.
Description: adverse respiratory events were defined as the occurrence of one or more clinical features of respiratory depression, including an oxygen saturation <91%, a change in baseline ETCO2 of >10 mm HG, or a loss of ETCO2 waveform, associated with the occurrence of any supportive airway maneuvers, including the use of a bag-valve mask apparatus, airway repositioning, the use of an oral or nasal airway to improve ventilation, or any stimulation to induce respirations.
Arm/Group | Moderate Procedural Sedation | Deep Procedural Sedation
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 21/54 | 24/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Procedural Sedation (N=54) | Deep Procedural Sedation (N=53)
adverse respiratory event (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 24 (40) — The occurrence of one or more clinical features of respiratory depression, defined as any oxygen saturation <91%, a change in baseline ETCO2 of >10mmhg, or a loss of ETCO2 waveform, associated with a supportive airway maneuver

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT02404610/Prot_SAP_000.pdf